CLINICAL TRIAL: NCT00120211
Title: Phase III Trial of Five Versus Six Fractions Per Week for Head and Neck Cancer
Brief Title: Trial of Five Versus Six Fractions Per Week for Head and Neck Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: International Atomic Energy Agency (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E33018
Record Dates: First submitted 2005-07-08; First posted 2005-07-15 (Estimated); Last update posted 2011-10-13 (Estimated); Status verified 2011-10

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms

ARMS (2):
- Radiotherapy: 6 Fractions (Experimental)
  Interventions: Radiation: Accelerated Radiotherapy Fractionation
- Radiotherapy: 5 fractions (Active Comparator)
  Interventions: Radiation: Accelerated Radiotherapy Fractionation

INTERVENTIONS:
Radiation: Accelerated Radiotherapy Fractionation — Radiation Therapy 6 fractions per week
  Arms: Radiotherapy: 6 Fractions
Radiation: Accelerated Radiotherapy Fractionation — Radiotherapy 5 fractions per week
  Arms: Radiotherapy: 5 fractions

SUMMARY:
This trial compares the use of 6 fractions versus the standard 5 fractions of radiotherapy used in the treatment of head and neck cancer.

DETAILED DESCRIPTION:
The purpose of this trial is to study the clinical effects of increasing the weekly fraction number for locally advanced head and neck cancers by a multi-institutional prospective randomised trial. The primary endpoint is to clarify whether a six fraction per week protocol has a greater effect on the survival, as compared to the conventional five fraction per week protocol.

ELIGIBILITY:
Inclusion Criteria:

* Head and Neck Cancer

Exclusion Criteria:

* Unable to give an informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 855 (Actual)
Dates: Start 1998-09; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Three Years Loco-regional Control | 3 years

SECONDARY OUTCOMES:
Disease-specific Survival | 8 years
Overall Survival | 8 years
Acute Adverse Effects
Late Adverse Effects | 8 years

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Rosenblatt, M.D., Study Director — International Atomic Energy Agency (IAEA)

REFERENCES:
- [Derived] Overgaard J, Mohanti BK, Begum N, Ali R, Agarwal JP, Kuddu M, Bhasker S, Tatsuzaki H, Grau C. Five versus six fractions of radiotherapy per week for squamous-cell carcinoma of the head and neck (IAEA-ACC study): a randomised, multicentre trial. Lancet Oncol. 2010 Jun;11(6):553-60. doi: 10.1016/S1470-2045(10)70072-3. Epub 2010 Apr 8. PMID 20382075
- See also: International Atomic Energy Agency, Research Contracts Administration — http://www.iaea.org